CLINICAL TRIAL: NCT02979145
Title: Development of the Charcot-Marie-Tooth Disease Infant Scale (CMTInfS) for Infants With CMT
Brief Title: Charcot-Marie-Tooth Disease (CMT) Infant Scale (INC-6611)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sydney Children's Hospitals Network (Other)
Collaborators: University of Iowa (Other); Children's Hospital of Philadelphia (Other); University of Pennsylvania (Other); University of Rochester (Other); National Hospital of Neurology and Neurosurgery (Unknown); Dubowitz Neuromuscular Centre (Other); University of Miami (Other); Carlo Besta Neurological Institute (Other); Johns Hopkins University (Other); Vanderbilt University (Other); University of Washington (Other); Nemours Children's Hospital (Other); National Institutes of Health (NIH) (NIH); Stanford University (Other); Cedars-Sinai Medical Center (Other); Harvard/Massachusetts General Hospital (Unknown); University of Michigan (Other); University of Minnesota (Other); University of Utah (Other); University of Connecticut (Other); Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Joshua Burns, Professor of Allied Health (Paediatrics), Sydney Children's Hospitals Network
Other Study IDs: 6611
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Charcot-Marie-Tooth Disease
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients with CMT: Two groups of patients will be included: Group 1 (Definitive): Children with known CMT where genetic testing confirms the diagnosis, or children with a clinical diagnosis including electrophysiology confirming the presence of CMT and a corresponding family history where a first or second degree relative has a genetic diagnosis; or Group 2 (At risk): A clinical diagnosis of CMT awaiting genetic testing or confirmatory electrophysiology and evidence of a genetic diagnosis in a first or second degree relative; or individuals identified as being at risk of a CMT diagnosis (prodromal patients), without the onset of signs or symptoms.
  Interventions: Other: No intervention involved
- Controls: Healthy controls will be included from unaffected family members or friends accompanying patients at INC sites. Healthy controls are defined as boys and girls aged 0-≤4 years without a diagnosis of CMT or any of the other study exclusion criteria.
  Interventions: Other: No intervention involved

INTERVENTIONS:
Other: No intervention involved

SUMMARY:
The purpose of this study is to develop and validate a clinical outcome measure to evaluate disability and disease progression of children 3 years of age and younger (infants and toddlers) with various types of Charcot-Marie-Tooth disease (CMT).

DETAILED DESCRIPTION:
Most forms of CMT begin in childhood and progress throughout a person's lifetime. Current research suggests that treatment to slow disease progression may be most effective if introduced early in a patient's life before muscle weakness and sensation loss develop, as it may be easier to slow disease progression than to reverse disability that is already in place. Clinical outcome measures have been developed for adults (CMT Neuropathy Score) and for children 3 years of age and older (CMT Pediatric Scale). However, no CMT-specific clinical outcome measure currently exists to measure disease severity or progression in children from birth to 3 years of age. It is the goal of this study to develop and validate the CMT Infant Scale (CMTInfS) to meet this need.

ELIGIBILITY:
Inclusion Criteria (patients with CMT):

* Patient is ≤4 years of age
* Parent(s) or guardians have agreed for the child to take part in the study and have signed an informed consent form.
* Patient has known or probable inherited neuropathy
* Patient participates in the INC Natural History Study (INC 6601)

Inclusion Criteria (controls):

* Participant is ≤4 years of age
* Parent(s) or guardians have agreed for the child to take part in the study and have signed an informed consent form.
* Participant does NOT have an inherited neuropathy as determined by the investigator
* Participant is an unaffected friend or family member of a patient with CMT (patient does not have to be included in the study)

Exclusion Criteria (patients with CMT):

* Patient has a known condition of acquired neuropathy including toxic (e.g. medication related), metabolic (e.g. diabetic), immune mediated or inflammatory (AIDP or CIDP) neuropathies, a neuropathy related to leukodystrophy, or a congenital muscular dystrophy.
* Patient has a severe general medical condition, as determined by the site Principal Investigator.
* Patient has known normal nerve conductions of upper and lower limbs. This will be considered as exclusion criteria because it documents that the child does not have a large-fibre neuropathy. However, patients will not be required to have nerve conduction studies (NCS) or electromyography (EMG).

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients who are 4 years of age and under who are also enrolled in the 6601 study and have performed all tasks to complete the CMTInfant Scale will be recruited for participation. Participation entails allow the information collected in the 6601 study be used for validation in the current study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
CMT Infant Scale Part 1 | 1 year
  The CMT Infant Scale physical assessment
The CMT Infant Scale Part 2 | 1 year
  The CMT Infant Scale lower limb and gross motor items
The CMT Infant Scale Part 3 | 1 year
  The CMT Infant Scale upper limb and fine motor items

SECONDARY OUTCOMES:
Evaluate CMT Infant Scale (CMTInfS) in CMT natural history study | 6 months - 1 year
  The sections of the CMT Infant Scale which are found to be clinically/functionally useful after one year of analysis will be carried forward for all infant patients every 6 months to one year.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - University of Iowa Health Care, Iowa City, Iowa
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- The Children's Hospital at Westmead, Sydney, New South Wales, Australia
- C. Besta Neurological Institute, Milan, Italy

REFERENCES:
- See also: 6611: Charcot-Marie-Tooth disease Infant Scale Recruitment Website — https://www.rarediseasesnetwork.org/cms/inc/6611